CLINICAL TRIAL: NCT06295991
Title: The Effect of Lycra Garment on Balance and Respiratory Functions in Spastic Diplegic Cerebral Palsy Individuals With Scoliosis
Brief Title: The Effect of Lycra Garment on Spastic Diplegic Cerebral Palsy Individuals With Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatih Çelik, PhD(s), Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2023/005
Record Dates: First submitted 2023-11-22; First posted 2024-03-06 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Balanced; Rearrangement; Respiratory Function Test
Keywords: lycra garment; diplegic cerebral palsy; balance; respiratory function; scoliosis
MeSH Terms: conditions — Cerebral Palsy; Respiratory Aspiration; Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): wearing lycra garment
  Interventions: Device: Lycra garment
- control group (Placebo Comparator): wearing non-lycra garment
  Interventions: Device: Lycra garment

INTERVENTIONS:
Device: Lycra garment — Investigation of the effect on balance and respiratory functions by using specially produced lycra garments for 6 hours a day for 16 weeks

SUMMARY:
The primary aim of this study was to investigate the effects of lycra clothing on balance and respiratory functions in individuals with cerebral palsy with scoliosis, and the secondary aim was to investigate the effects of lycra clothing on motor function, activity limitation and quality of life in these individuals.

DETAILED DESCRIPTION:
H.3. Scope: Cerebral palsy (CP) is defined as a permanent, non-progressive abnormality in motor function as a result of injury to the developing brain. Spinal deformity is a common musculoskeletal problem in individuals with cerebral palsy. There is a strong link between CP and the development of scoliosis. It is estimated that 21% to 64% of individuals with CP have scoliosis. It has also been suggested that there is an inverse relationship between the development of scoliosis and ambulation and the least mobile individuals are at the greatest risk. Gu et al. suggested that age was the most important risk factor, but they did not find a relationship between the height and weight of children and curve progression.

Two different scoliotic curve patterns have been defined in individuals with CP. Group-I curves can be considered as double curves with thoracic and lumbar components and occur most commonly in individuals who can walk with minimal pelvic obliquity (7). Group-II curves are single curves in the thoracic or lumbar spine and are larger. They are more common in quadriplegic individuals and almost all of them have marked pelvic obliquity.

The aim of non-surgical scoliosis treatment in CP is to improve sitting control and to reduce or change curve progression without the need for surgical intervention. Historical reports show that the use of supportive bracing in children with CP is poorly tolerated and ineffective. There is little evidence for the use of modern bracing techniques. However, more recent studies suggest that braces improve sitting balance and trunk support, which leads to better control of the head and neck as well as better use of the upper limbs as they do not need to support the trunk in a sitting position. Evidence regarding the use of orthosis to prevent scoliotic curve progression is mixed. Some authors have suggested that bracing may slow curve progression, especially in young individuals with curves less than 40 degrees.

In individuals with scoliosis, vertebral verticalisation due to deformity changes the position of the body centre of mass line, which may adversely affect postural balance and stabilisation. In addition, force imbalance between the spinal muscles may cause postural oscillations.

Impaired respiratory function, which is frequently observed in adolescents and adults with severe cerebral palsy (CP), is caused by underdevelopment of the upper chest wall. This underdevelopment prevents chest expansion and may cause rapid and paradoxical breathing patterns. Gravitational forces interact with forces generated from muscle contractions to facilitate the musculoskeletal development of an infant's thorax. The weak musculature of a young child with CP often cannot optimally balance gravitational forces and chest development is adversely affected. The incidence of scoliosis in CP and atypical chest wall structure and function are interrelated. Therefore, individuals with CP and scoliosis are likely to be adversely affected in respiratory functions both due to CP and scoliosis.

Method: Study Type and Participants This study, which is planned as a cross-sectional study, aims to include 24 volunteers aged 10-18 years with CP diagnosed with scoliosis.

Volunteers who agree to participate in the study will be divided into two groups (lycra clothing group/placebo group) by stratified randomisation method according to age and gender. Only individuals with diplegic type CP will be included in the study. After randomisation, the individuals in the lycra clothing group will be subjected to the assessments described below three times in total, once before wearing lycra clothing prepared with special measurements, once after 8 weeks of clothing use and once again after 16 weeks, without clothing. The individuals in the placebo group will be evaluated at the beginning, 8th week and 16th week in the same order by taking special measurements and using clothes prepared in the colour of lycra clothes but not compressing the body, that is, from fabric that does not have lycra properties. For 16 weeks, individuals will be provided to wear the determined clothes for 6 hours a day.

The fabric of the lycra clothing to be used in the study is an elastic fabric woven from fibres called elastane. The fabric to be used will be selected from 100% lycra woven fabric. In non-lycra clothes, completely cotton fabric will be used. In both clothing groups, measurements will be taken from the individual and for lycra clothes, according to the structure of scoliosis, elastic bands will be applied from the convex side apex points and over the lateralised hip, supported by soft, antiallergic plastazote. Lycra-free clothes will be produced in the same structure as lycra clothes in terms of appearance and colour, but the fabric to be used will be completely cotton, non-elastic and wide enough not to cover the body.

In addition to the physiotherapy programmes applied for 40 minutes 2 days a week, a scoliosis-specific exercise programme will be applied by the co-researcher (Fatih Çelik) for 20 minutes after each physiotherapy programme. The family will be asked to keep a diary for clothing care and use and will be regularly checked by the researcher during the scoliosis exercise programme to be applied in addition to physiotherapy sessions. The evaluations will be made by the co-researcher (Kamil Yılmaz) who does not know which individual wears which clothes and blinding will be applied.

Inclusion criteria (for study and control group) Being diagnosed with spastic diplegic CP Being diagnosed with scoliosis, To be between the ages of ten and eighteen, Being at I-II-III level according to GMFCS classification, Not having undergone scoliosis surgery, Cobb angle to be between 10-40 degrees, Receiving physiotherapy appropriate to the functional status for at least 6 months.

Exclusion criteria (for study and control group) Psychiatric disorders, Having a communication problem at a level that cannot adapt to the physiotherapist's instructions, To have undergone scoliosis surgery, Having uncontrolled epilepsy.

Assessments; Firstly, demographic information such as age, height, body weight and gender will be obtained.

The degree of spasticity will be determined with the modified ashworth scale and recorded.

Balance Assessment Posturography is a test method used to assess balance disorders. This test aims to objectively measure a person's balance control, body posture and movements. Posturography is usually performed on a balance platform. This platform is a surface equipped with pressure sensors. During the test, the person places their feet on the platform and performs various balance tasks. Sensors detect the distribution of the person's feet and body weight on the platform and analyse this information by transmitting it to a computer.

Assessment of Respiratory Functions Respiratory functions of the individuals will be measured with a spirometer using the spirometric measurement method whose validity and reliability has been proven by Finkelstein et al.

Motor Function Assessment For gross motor function assessment, the Gross Motor Function Measure (GMFM-66) developed by Palisano et al. which has validity and reliability in individuals with cerebral palsy aged 5-18 years will be used.

Functional Independence Assessment Functional Independence Measure (FIM), whose validity and reliability have been proven for both adolescents and adults, will be used.

Assessment of Activity Restriction Activity limitation will be evaluated with the ACTIVLIM questionnaire developed by Vandervelde et al. for use in adults and children.

Quality of Life Assessment The disease-related quality of life of the individuals included in the study will be evaluated with the Scoliosis Research Society 22nd Form (SRS 22r) scale developed by Alanay A. et al.

Posture Assessment Posture will be evaluated using the POTSI (posterior trunk symetry index) index. Its validity in scoliosis has been demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with spastic diplegic CP
* Being diagnosed with scoliosis,
* To be between the ages of ten and eighteen,
* Being at I-II-III level according to GMFCS classification (18),
* Not having undergone scoliosis surgery,
* Cobb angle to be between 10-40 degrees,
* To be receiving physiotherapy appropriate to the functional status for at least 6 months.

Exclusion Criteria:

* Psychiatric disorders,
* Having a communication problem at a level that cannot adapt to the physiotherapist's instructions,
* To have undergone scoliosis surgery,
* Uncontrolled epilepsy.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Balance parameters | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Measurement of balance control, body posture and body movement parameters using posturography
Respiratory functions | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Measurement of respiratory functions like as FEV1, FVC, VC, PEF, FEV1/FVC parameters with sipirometer
Respiratory muscle strength measurement | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Measurement of respiratory muscle strength as MIP/MEP parameters with Respiratory Pressure Meter (RPM)

SECONDARY OUTCOMES:
Gross motor function measurement | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Measurement of gross motor functions with "Gross Motor Function Measure-66 form"
Functional independence assessment | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Assessment of functional independence with "Functional Independence Measure (FIM)"
Assessment of activity restriction | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Evaluation of activity restriction with "AKTIVLIM" form
Quality of life assessment | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Assessment of quality of life with "SRS-22" form
Assessment of posture | At the beginning, at the end of the eighth week and at the end of the sixteenth week
  Postural assessment with "POTSI (posterior trunk symetry index)" index

CONTACTS AND LOCATIONS:
Overall Officials: İpek Gürbüz, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Fizyo Omurga, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Balmer GA, MacEwen GD. The incidence and treatment of scoliosis in cerebral palsy. J Bone Joint Surg Br. 1970 Feb;52(1):134-7. No abstract available. PMID 5436198
- [Background] Madigan RR, Wallace SL. Scoliosis in the institutionalized cerebral palsy population. Spine (Phila Pa 1976). 1981 Nov-Dec;6(6):583-90. doi: 10.1097/00007632-198111000-00009. PMID 7336281
- [Background] Persson-Bunke M, Hagglund G, Lauge-Pedersen H, Wagner P, Westbom L. Scoliosis in a total population of children with cerebral palsy. Spine (Phila Pa 1976). 2012 May 20;37(12):E708-13. doi: 10.1097/BRS.0b013e318246a962. PMID 22218299
- [Background] Saito N, Ebara S, Ohotsuka K, Kumeta H, Takaoka K. Natural history of scoliosis in spastic cerebral palsy. Lancet. 1998 Jun 6;351(9117):1687-92. doi: 10.1016/S0140-6736(98)01302-6. PMID 9734885
- [Background] Gu Y, Shelton JE, Ketchum JM, Cifu DX, Palmer D, Sparkman A, Jermer-Gu MK, Mendigorin M. Natural history of scoliosis in nonambulatory spastic tetraplegic cerebral palsy. PM R. 2011 Jan;3(1):27-32. doi: 10.1016/j.pmrj.2010.09.015. PMID 21257130
- [Background] Lonstein JE, Akbarnia A. Operative treatment of spinal deformities in patients with cerebral palsy or mental retardation. An analysis of one hundred and seven cases. J Bone Joint Surg Am. 1983 Jan;65(1):43-55. No abstract available. PMID 6848534
- [Background] Terjesen T, Lange JE, Steen H. Treatment of scoliosis with spinal bracing in quadriplegic cerebral palsy. Dev Med Child Neurol. 2000 Jul;42(7):448-54. doi: 10.1017/s0012162200000840. PMID 10972416
- [Background] Miller A, Temple T, Miller F. Impact of orthoses on the rate of scoliosis progression in children with cerebral palsy. J Pediatr Orthop. 1996 May-Jun;16(3):332-5. doi: 10.1097/00004694-199605000-00007. PMID 8728632
- [Background] Olafsson Y, Saraste H, Al-Dabbagh Z. Brace treatment in neuromuscular spine deformity. J Pediatr Orthop. 1999 May-Jun;19(3):376-9. PMID 10344323
- [Background] Kubat O, Ovadia D. Frontal and sagittal imbalance in patients with adolescent idiopathic deformity. Ann Transl Med. 2020 Jan;8(2):29. doi: 10.21037/atm.2019.10.49. PMID 32055620
- [Background] de Santiago HA, Reis JG, Gomes MM, da Silva Herrero CF, Defino HL, de Abreu DC. The influence of vision and support base on balance during quiet standing in patients with adolescent idiopathic scoliosis before and after posterior spinal fusion. Spine J. 2013 Nov;13(11):1470-6. doi: 10.1016/j.spinee.2013.03.027. Epub 2013 Apr 25. PMID 23623510
- [Background] Massery M. Chest development as a component of normal motor development: implications of pediatric physical therapists. Pediatr Phys Ther. 1991;3(1):3-8.
- [Background] Moerchen V. Respiration and motor development: a systems perspective. Neurol Rep. 1994;18:8-10.
- [Background] Kotwicki T, Jozwiak M. Conservative management of neuromuscular scoliosis: personal experience and review of literature. Disabil Rehabil. 2008;30(10):792-8. doi: 10.1080/09638280801889584. PMID 18432437
- [Background] Banta JV, Drummond DS, Ferguson RL. The treatment of neuromuscular scoliosis. Instr Course Lect. 1999;48:551-62. No abstract available. PMID 10098083
- [Background] Rennie DJ, Attfield SF, Morton RE, Polak FJ, Nicholson J. An evaluation of lycra garments in the lower limb using 3-D gait analysis and functional assessment (PEDI). Gait Posture. 2000 Sep;12(1):1-6. doi: 10.1016/s0966-6362(00)00066-7. PMID 10996291
- [Background] Bodkin AW, Robinson C, Perales FP. Reliability and validity of the gross motor function classification system for cerebral palsy. Pediatr Phys Ther. 2003 Winter;15(4):247-52. doi: 10.1097/01.PEP.0000096384.19136.02. PMID 17057460
- [Background] Mutlu A, Livanelioglu A, Gunel MK. Reliability of Ashworth and Modified Ashworth scales in children with spastic cerebral palsy. BMC Musculoskelet Disord. 2008 Apr 10;9:44. doi: 10.1186/1471-2474-9-44. PMID 18402701
- [Background] Visser JE, Carpenter MG, van der Kooij H, Bloem BR. The clinical utility of posturography. Clin Neurophysiol. 2008 Nov;119(11):2424-36. doi: 10.1016/j.clinph.2008.07.220. Epub 2008 Sep 12. PMID 18789756
- [Background] Finkelstein SM, Lindgren B, Prasad B, Snyder M, Edin C, Wielinski C, Hertz M. Reliability and validity of spirometry measurements in a paperless home monitoring diary program for lung transplantation. Heart Lung. 1993 Nov-Dec;22(6):523-33. PMID 8288456
- [Background] Palisano RJ, Rosenbaum P, Bartlett D, Livingston MH. Content validity of the expanded and revised Gross Motor Function Classification System. Dev Med Child Neurol. 2008 Oct;50(10):744-50. doi: 10.1111/j.1469-8749.2008.03089.x. PMID 18834387
- [Background] Ataç, T. (2020). Serebral Palsili Çocuklarda Kaba Motor Fonksiyon Ölçütünün Uzun (Kmfö-88) ve Kısa (Kmfö-66) Formunun Türkçeye Uyarlanması, Güvenilirlik ve Geçerliliğinin Araştırılması ve Klinik Tiplere Göre İncelenmesi.
- [Background] Kidd D, Stewart G, Baldry J, Johnson J, Rossiter D, Petruckevitch A, Thompson AJ. The Functional Independence Measure: a comparative validity and reliability study. Disabil Rehabil. 1995 Jan;17(1):10-4. doi: 10.3109/09638289509166622. PMID 7858276
- [Background] Alanay A, Cil A, Berk H, Acaroglu RE, Yazici M, Akcali O, Kosay C, Genc Y, Surat A. Reliability and validity of adapted Turkish Version of Scoliosis Research Society-22 (SRS-22) questionnaire. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2464-8. doi: 10.1097/01.brs.0000184366.71761.84. PMID 16261127
- [Background] Suzuki, N., et al. Analysis of posterior trunk symmetry index (POTSI) in scoliosis. Part 1. Research into spinal deformities, 1999, IOS Press: 81-84.
- [Background] Vandervelde L, Van den Bergh PY, Goemans N, Thonnard JL. ACTIVLIM: a Rasch-built measure of activity limitations in children and adults with neuromuscular disorders. Neuromuscul Disord. 2007 Jun;17(6):459-69. doi: 10.1016/j.nmd.2007.02.013. Epub 2007 Apr 11. PMID 17433675